CLINICAL TRIAL: NCT05254340
Title: A Novel Approach to Measuring Intestinal Production of Short Chain Fatty Acids: A Proof-of-concept Healthy Volunteer Study
Brief Title: Healthy Volunteer Short Chain Fatty Acid Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study physician left the university
Sponsor: Indiana University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Huiping Xu, Associate Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010116953; K23DK122015 (NIH)
Record Dates: First submitted 2021-10-07; First posted 2022-02-24 (Actual); Results first posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Healthy
Keywords: bile acid; inulin; microbiota
MeSH Terms: interventions — Inulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteers (Experimental): Adults ages 18-75 years with no prior history of gastrointestinal diseases or symptoms.
  Interventions: Dietary Supplement: Inulin

INTERVENTIONS:
Dietary Supplement: Inulin — Inulin ingestion is not being used to diagnose, treat, or prevent irritable bowel syndrome. Inulin is being used to study an individual's ability to ferment dietary fiber.

SUMMARY:
The purpose of this study is to evaluate the production of short chain fatty acids (fatty acids are part of your diet) in stool through the measurement of fecal inulin after a one-time ingestion of 10-gram dose of inulin among healthy adult volunteers.

DETAILED DESCRIPTION:
The Study involves 2 visits and will include 3 types of subjects. Any healthy adult between the ages of 18 and 75 with no prior history of GI disease or symptoms is eligible to participate in the study.

Visit 1 (Day 1) - Screening Visit and Informed Consent At this Visit volunteers will do the following

* Volunteers will be asked to read and sign the informed consent after all questions about the study have been answered. This is a screening visit, and we may determine that the volunteers ineligible to continue to participate in the study.
* Volunteers will have medical history taken including demographics, symptoms and history of illness.
* Volunteers will be asked about the medications.
* A physical exam will be performed by the physician.
* Vital signs will be measured.
* Volunteers will be scheduled for study-days and will fill out a bowel disease questionnaire (BDQ).
* Volunteers will be provided instructions for collection, storage, and transportation of stool for your next visit.
* Volunteers will be provided a kit for stool collection, storage, and transportation.
* Volunteers will be provided a bowel pattern diary to record bowel symptoms over the course of the study.
* Volunteers will also be provided with 10-gram inulin powder supplement and will be required to consume the inulin before 9 am on Day 2.

Day 2 (at home):

* Day 2 reflects the first day of active study. Day 2 may occur anytime up to 30 days after Day 1. This will depend whether the volunteers need to stop any medications or on the day they are able to return for the final visit.
* Volunteers will have to consume the inulin supplement before 9 am on Day 2. The first 24-hour stool collection will begin starting at 7 am on Day 2 and will continue until 7 am on Day 3.
* All collected stool should be stored as per instructions provided on Day 1 (screening visit).
* Volunteers will be asked to record bowel symptoms using the bowel diary card and dietary intake data for four days from Day 2 through Day 5 by using diaries (diet information may be recorded using either the paper diaries that are provided or the web-based Automated Self-Administered Dietary Assessment Tool (https://epi.grants.cancer.gov/asa24/).

Day 3 to 4 (at home) - The second 24-hour stool collection will begin starting at 7 am on Day 3 and continue until 7 am Day 4. Volunteers will record the diet for Day 3 to 4 as "Day 3 Diet" and will record bowel symptoms using a Bowel Diary Card.

Day 4 to 5 (at home)- Volunteers will start third 24-hour stool collection at 7 am on Day 4 and continue until 7 am Day 5. The diet for Day 4 to 5 should be recorded as "Day 4 Diet." Volunteers will record the bowel symptoms using a Bowel Diary Card.

Day 5 to 6 (at home)- The fourth 24-hour stool collection begins at 7 am on Day 5 and continue until 7 am Day 6. Volunteers will record the diet for Day 5 to 6 as "Day 5 Diet" and will record bowel symptoms using a Bowel Diary Card.

Visit 2 (Day 6) - End of study: Volunteers will return the refrigerated stool specimens, bowel diaries and dietary intake diaries to the study team. Diaries may also be returned by mail, fax, or by electronic submission. For the diet diaries, volunteers will have the option to complete paper diaries or the Automated Self-Administered Dietary Assessment. Volunteers' participation in the study will end after this visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults ages 18-75 years with no prior history of GI disease or symptoms.
* Participants should be on a stable and consistent diet regimen and should not be following an extreme diet intervention such as gluten-free or a low fermentable oligo-, di-, monosaccharides, and polyols diet (FODMAP) diet at the time of study participation

Exclusion Criteria:

* History of microscopic colitis, inflammatory bowel disease, celiac disease, visceral cancer, chronic infectious disease, immunodeficiency, uncontrolled thyroid disease, history of liver disease or history of elevated aspartate transaminase/alanine transaminase > 2.0x the upper limit of normal
* Prior therapy of the abdomen or abdominal surgeries with the exception of appendectomy or cholecystectomy > 6 months prior to study initiation
* Ingestion of any prescription, over the counter, or herbal medications which can affect study interpretation within 6 months of study initiation for asymptomatic volunteers. Rescue therapy to facilitate stool collection will be permitted where needed.
* Any females who are pregnant or breast-feeding
* Antibiotic usage within 3 months prior to study participation
* Prebiotic or probiotic usage within the 2 weeks prior to study initiation
* Inulin usage within the 2 weeks prior to study initiation
* Use of tobacco products within the past 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Volunteers: Adults ages 18-75 years with no prior history of gastrointestinal diseases or symptoms.
  Inulin: Inulin ingestion is not being used to diagnose, treat, or prevent irritable bowel syndrome. Inulin is being used to study an individual's ability to ferment dietary fiber.
  All subjects received the same intervention so we report them as one group with no stratification.
Period: Overall Study
Arm/Group | Healthy Volunteers
Started | 29
Completed | 22
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex was not reported for 3 subjects
  Participants
    number analyzed (Participants) | 26
    Female | 13
    Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 13
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Fecal Inulin
Description: Fecal inulin content will be measured using short acid hydrolysis and high-performance liquid chromatography
Time Frame: 4 days
Population: Fecal inulin was missing for 7 subjects who completed the study
Measure: Median (Inter-Quartile Range); unit: ug/1 mL extract
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 15
ug/1 mL extract | 45.2 [34.6 to 58.6]

2. Primary Outcome: Total Fecal Short Chain Fatty Acids
Description: Stool samples will be collected for measurement of measurement of short chain fatty acids (mmol/kg) by liquid chromatography-mass spectrometry
Time Frame: 4 days
Population: One subject completing the study had missing data on short chain fatty acids
Measure: Median (Inter-Quartile Range); unit: mmol/kg
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 21
mmol/kg | 207.4 [159.7 to 375.5]

3. Primary Outcome: Individual Fecal Short Chain Fatty Acids
Description: as for outcome 2
Time Frame: 4 days
Population: One subject completing the study had missing data on short chain fatty acids
Measure: Median (Inter-Quartile Range); unit: mmol/kg
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 21
mmol/kg
  Acetic Acid | 111.5 [99.4 to 279.7]
  Priopionic Acid | 37.3 [26.8 to 63.5]
  Butyric Acid | 51 [25.1 to 60.3]

4. Secondary Outcome: Bowel Frequency
Description: Stool characteristics will be measured using a 4 day bowel diary (stool frequency, stool form, ease of passage). Bowel frequency indicates the total number of bowel movements in 4 days.
Time Frame: 4 days
Population: 5 subjects did not complete the bowel diary, resulting in missing data.
Measure: Median (Inter-Quartile Range); unit: Number of bowel movements
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 17
Number of bowel movements | 4 [4 to 4]

5. Secondary Outcome: Dietary Intake
Description: Baseline dietary intake will be measured using an automated self-administered dietary assessment tool
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: kcal
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 18
kcal | 2065.9 [1415.6 to 2666.1]

6. Secondary Outcome: Bowel Symptoms
Description: Stool characteristics will be measured using a 4 day bowel diary (stool frequency, stool form, ease of passage). Stool form is on a scale from 1 to 7, where 1=hard lumps, 2=lumps sausage, 3=cracked sausage, 4=normal, 5=soft lumps, 6=mushy, 7=watery, summarized on the level of bowel movements. Ease of passage is on a scale from 1 to 7, where 1=manual disimpaction, 2=enema needed, 3=straining needed, 4=normal, 5=urgent without pain, 6=urgent with pain, 7=incontinent, also summarized on the level of bowel movements.
Time Frame: 4 days
Measure: Median (Inter-Quartile Range); unit: units on a scale
Units Other Than Participants: Bowel movements
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 17
Number analyzed (Bowel movements) | 65
units on a scale
  Stool form | 4 [3 to 5]
  Ease of passage | 4 [4 to 4]

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT05254340/Prot_SAP_000.pdf